CLINICAL TRIAL: NCT04740203
Title: Clinical Trial for the Safety and Efficacy of Sequential CD19 and CD22 CAR-T Therapy for Adult Patients With Newly Diagnosed Ph Chromosome Negative B-cell Acute Lymphoblastic Leukemia
Brief Title: Sequential CD19 and CD22 CAR-T Therapy for Newly Diagnosed Ph- B-ALL
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang University (Other)
Collaborators: Yake Biotechnology Ltd. (Industry)
Responsible Party: Principal Investigator, He Huang, Professor, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD19-005
Record Dates: First submitted 2021-01-31; First posted 2021-02-05 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: B-Cell Acute Lymphoblastic Leukemia, Adult
Keywords: CD19 CAR-T; CD22 CAR-T; Ph Chromosome Negative; B-ALL; Newly diagnosed
MeSH Terms: conditions — Burkitt Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T therapy (Experimental): Administration of CD19 and CD22 CAR T-cells
  Interventions: Drug: CAR-T cells targeting CD19 and CD22

INTERVENTIONS:
Drug: CAR-T cells targeting CD19 and CD22 — Each subject receives sequential CD19 and CD22 CAR-T cells by intravenous infusion

SUMMARY:
Clinical Trial for the Safety and Efficacy of Sequential CD19 and CD22 CAR-T Therapy for Adult Patients With Newly Diagnosed Ph Chromosome Negative B-cell Acute Lymphoblastic Leukemia

DETAILED DESCRIPTION:
This is a prospective, single arm study. To evaluate the safety and efficacy of sequential CD19 and CD22 CAR-T cells in the treatment of adult newly diagnosed Ph chromosome negative B-cell acute lymphoblastic leukemia. The main endpoints were dose limiting toxicity (DLT) and incidence of adverse events (TEAEs).

ELIGIBILITY:
Inclusion Criteria:

* Age≥15 years old
* Newly diagnosed B-cell acute lymphoblastic leukemia according to the 2016 WHO classification
* The immunophenotype of leukemia cells were CD19 and CD22 positive
* Ph- or Ph- like negative
* Anticipated survival time more than 12 weeks;
* Those who voluntarily participated in this trial and provided informed consent.

Exclusion Criteria:

* History of craniocerebral trauma, conscious disturbance, epilepsy, cerebrovascular ischemia, and cerebrovascular hemorrhagic diseases;
* Electrocardiogram shows prolonged QT interval, severe heart diseases such as severe arrhythmia in the past;
* Pregnant (or lactating) women;
* Patients with severe active infections (excluding simple urinary tract infection and bacterial pharyngitis);
* Active infection of hepatitis B virus or hepatitis C virus;
* Concurrent therapy with systemic steroids within 2 weeks prior to screening, except for the patients recently or currently receiving inhaled steroids;
* Previously treated with any CAR-T cell product or other genetically-modified T cell therapies;
* Creatinine>2.5mg/dl, or ALT / AST > 3 times of normal amounts, or bilirubin>2.0 mg/dl;
* Other uncontrolled diseases that were not suitable for this trial;
* Patients with HIV infection;
* Any situations that the investigator believes may increase the risk of patients or interfere with the results of study.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-01-31 (Estimated); Primary Completion 2024-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Baseline up to 28 days after CAR-T cells infusion
  Adverse events assessed according to NCI-CTCAE v5.0 criteria
Incidence of treatment-emergent adverse events (TEAEs) | Up to 2 years after CAR-T cells infusion
  Incidence of treatment-emergent adverse events [Safety and Tolerability]

SECONDARY OUTCOMES:
Complete Remission Rate | up to 28 days after CAR-T cells infusion
  Complete Remission Rate after CAR-T cell therapy
Overall survival (OS) | Up to 2 years after CD19 CAR-T cells infusion
  From the first infusion of CD19 CAR-T cells to death or the last visit
Leukemia-free survival (LFS) | Up to 2 years after CD19 CAR-T cells infusion
  From the complete remission to the occurrence of any event, including death, relapse (any one occurs first), and the last visit
Quality of life | At Baseline, Month 1, 3, 6, 9 and 12
  Assessment using European Organisation for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) scale [For item1-28: max score: 112, min score: 28, higher scores mean a better outcome; for item 28-29: max score: 14, min score: 2, higher scores mean a worse outcome] to measure Quality of life at Baseline, Month 1, 3, 6, 9 and 12

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No